CLINICAL TRIAL: NCT00199459
Title: Urinary Proteomic Profiling Using ProteinChip SELDI-TOF-MS: A Potential Means of Identifying Protein Biomarkers of Urinary Stone Formers
Brief Title: Proteomic Study of Urinary Stone Disease
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); University of Western Ontario, Canada (Other)
Responsible Party: Dr. John D. Denstedt, St. Joseph's Health Care London
Other Study IDs: R-04-481; PSI 04-041
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Urinary Calculi; Hyperoxaluria; Calculi
Keywords: calculi; proteomics
MeSH Terms: conditions — Urinary Calculi; Hyperoxaluria; Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Urinary protein levels are not routinely measured in stone patients while there is strong evidence that proteins play a role in the etiology of stones. The purpose of this study is to examine the urinary and serum proteins of stone formers compared to healthy subjects utilizing the high throughput method, Surface Enhanced Laser Desorption/Ionization (SELDI). We hypothesize that there is a unique set of proteins expressed in serum and urine in stone patients that can be detected by SELDI. Ultimately, this will better our understanding of stone disease and help develop new prevention strategies.

DETAILED DESCRIPTION:
Urinary stone disease affects 10% of the Canadian population during their lifetime and approximately half of these patients will have another episode within ten years. Currently, patients undergo metabolic testing (serum and 24 hour urine tests) to identify modifiable risk factors; however, no modifiable risk factors are identified in many patients, yet they continue to form stones. New techniques must be developed to identify stone patients at risk for future recurrences and ultimately to develop more specific prevention strategies.

Urinary protein levels are not routinely measured in stone patients while there is strong evidence that proteins play a role in the etiology of stones. The purpose of this study is to examine the urinary and serum proteins of stone formers compared to healthy subjects utilizing the high throughput method, Surface Enhanced Laser Desorption/Ionization (SELDI). We hypothesize that there is a unique set of proteins expressed in serum and urine in stone patients that can be detected by SELDI. Once a protein is identified as a biomarker, a specific assay similar to a quick and affordable dipstick test may be developed to identify those stone patients at risk of future stones. Ultimately, this will better our understanding of stone disease and help develop new prevention strategies.

Comparisons: protein profiles (serum/urine) of stone patients both during the presence of a stone and 6 weeks after they have passed it. comparison of stone profiles of stone patients with controls (non-forming stone patients).

ELIGIBILITY:
Inclusion Criteria:

* Controls:

  * Ages 18 to 65 years of age
  * No history of stone disease and no radiographical evidence of stone (as demonstrated by negative ultrasound)
  * No family history of stones
  * Healthy and no autoimmune or systemic disease that may affect renal function (see exclusion criteria)

Stone patients

* Ages 18 to 65 years of age
* Solitary stone of any size, in any location along the urinary tract (except lower renal calyceal stones and bladder stones)
* Radiology of any modality proving the existence of the stone (ultrasound, computed tomography, intravenous pyelogram, kidney-ureter-bladder x-ray)

Exclusion Criteria:

* ALL:

  * Pregnant females
  * Male patients treated for with benign prostate hyperplasia (BPH) (ongoing medical treatment or surgical intervention within 6 months)
  * Positive urine culture
  * Any cancer (excluding superficial skin, brain)
  * Chronic Recurrent urinary infections (prostate, cystitis, vaginosis/vaginitis)
  * Gross hematuria
  * Autoimmune disease that may affect renal function (eg Systemic lupus erythematosus)
  * Renal dysfunction or its common causes:
  * Diabetes
  * Uncontrolled hypertension (with concurrent microalbuminuria) (diastolic BP > 90 mmHg)
  * glomerulonephritis
  * Renal transplant
  * Genetic stone disease (e.g. Cystine stones, xanthinuria)
  * Medullary sponge kidney, or other renal anomalies such as horseshoe kidney
  * GI disorders: Inflammatory bowel disease, short bowel
  * Hypercalcemic disorders (hyperparathyroidism, sarcoidosis, Paget's disease)
  * Renal tubular acidosis
  * Immunodeficient patients e.g. HIV (indinavir stones)
  * Unable to provide informed consent
  * Anyone in the opinion of the investigator who would be inappropriate

Controls :

* In addition to criteria above.....
* persistent thiazide use
* Family history of stones (this will exclude any genetic factors since a positive family history increases the risk of urolithiasis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This observational study will compare stone formers meeting the inclusion criteria with a cohort of age and sex matched non-stone formers as controls.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Denstedt, MD, FRCSC, Principal Investigator — The University of Western Ontario (Professor)
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada